CLINICAL TRIAL: NCT01160445
Title: Phase II Study of Aldesleukin (IL-2) Following the Administration of Zanolimumab (Anti-CD4mAb) in Metastatic Melanoma and Metastatic Renal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated because we were not able to obtain the study drug.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100145; 10-C-0145
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Melanoma; Metastatic Renal Cancer
Keywords: Metastatic Melanoma; Metastatic Kidney Cancer; Clinical Performance; Tumor Regression; Toxicity
MeSH Terms: conditions — Melanoma; Kidney Neoplasms | interventions — zanolimumab; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD IL-2 + Zanolimumab - Melanoma (Experimental): Patients with metastatic melanoma Zanolimumab 14 mg/kg as an intravenous infusion weekly (+/- 3 days) for 9 weeks.
  Aldesleukin (IL-2) 720,000 IU/kg every 8 hours for a maximum of 15 doses.
  Interventions: Drug: Zanolimumab; Drug: Aldesleukin
- HD IL-2 + Zanolimumab - Renal Cell (Experimental): Patients with metastatic renal cancer Zanolimumab 14 mg/kg as an intravenous infusion weekly (+/- 3 days) for 9 weeks.
  Aldesleukin (IL-2) 720,000 IU/kg every 8 hours for a maximum of 15 doses.
  Interventions: Drug: Zanolimumab; Drug: Aldesleukin

INTERVENTIONS:
Drug: Zanolimumab — 14 mg/kg as an intravenous infusion weekly (+/- 3 days) for 9 weeks.
  Other Names: HuMax-CD4
Drug: Aldesleukin — 720,000 IU/kg every 8 hours for a maximum of 15 doses.
  Other Names: IL-2

SUMMARY:
Background:

* Aldesleukin (IL-2) is a drug that can help to shrink tumors in some patients with metastatic renal cancer and metastatic melanoma. It is possible that removing certain white blood cells (known as CD4 cells) before IL-2 treatment may improve the treatment effects.
* Zanolimumab is an antibody that works by destroying CD4 cells in the blood. Researchers are interested in determining whether zanolimumab can improve the results of IL-2 treatment if it is given before, during, and after IL-2 treatment. In addition, further research with zanolimumab may provide more information on how IL-2 treatment causes tumors to stop growing or shrink.

Objectives:

- To evaluate the effectiveness of IL-2 treatment in conjunction with zanolimumab in individuals with metastatic cancer.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with metastatic melanoma or metastatic kidney cancer.

Design:

* Eligible participants will be screened with a full physical examination and medical history, imaging studies, and blood samples, including leukapheresis, to remove a sample of white blood cells for testing purposes. Participants may also have a colonoscopy and biopsies if they have received previous treatments that have been known to cause colon damage.
* Participants will be treated with zanolimumab and IL-2 treatment for 9 weeks.
* Zanolimumab will be given on an outpatient basis during weeks 1 through 4, 6, 8, and 9. In weeks 5 and 7, participants will receive zanolimumab as an inpatient in addition to IL-2 therapy.
* Inpatient IL-2 treatment will be given during weeks 5 and 7. Up to 15 doses of IL-2 treatment will be given over a maximum of 5 days, followed by inpatient recovery time.
* During week 5, participants will have tumor imaging studies prior to receiving zanolimumab and IL-2 treatment.
* About 2 weeks after the treatment period, participants will return to the clinical center for a 2-day evaluation with a physical examination, imaging studies, and blood samples.
* Participants whose tumors have responded to treatment will be offered up to two additional courses of treatment, starting 6 to 8 weeks after the last IL-2 dose. Subsequent courses will be given exactly as described above in the initial course of treatment. Participants whose tumors do not respond to treatment will have follow-up evaluations as required by the study researchers.

DETAILED DESCRIPTION:
Background:

Zanolimumab is a human monoclonal antibody (mAb) that specifically recognizes CD4 protein expressed on a subset of T lymphocytes and on monocytes from humans, and non-human primates.

Ongoing clinical studies have identified a 14 mg/kg dose of zanolimumab weekly as a safe and efficacious dose. Toxicities of zanolimumab included headache, influenza-like illness, injection/infusion site reaction, nasopharyngitis, pyrexia, diarrhea, fatigue, and cytokine release syndrome at the time of infusion.

The current protocol is based on the hypothesis that transient elimination of CD4+ T-regulatory cells with zanolimumab will enhance the clinical effectiveness of aldesleukin (IL-2) administration by decreasing T-regulatory cell generation.

Objectives:

Primary objective:

Determine the ability of a combination of aldesleukin and zanolimumab (anti-CD4 mAb) administration to mediate tumor regression in patients with metastatic melanoma and metastatic kidney cancer.

Secondary objectives:

Determine the rate of depletion and repopulation of CD4+ cells.

Determine the toxicity of this treatment.

Determine the potential for pharmacokinetic interaction between zanolimumab and aldesleukin.

Eligibility:

Patients who are 18 years of age or older must have:

measurable metastatic melanoma or metastatic kidney cancer;

clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, or 1.

Patients may not have:

previously received high dose aldesleukin.

Design:

Patients will receive zanolimumab at a dose of 14 mg/kg as an intravenous (i.v.) infusion weekly for 9 weeks. After the fifth and seventh dose of zanolimumab, aldesleukin will administered as an i.v. bolus at a dose of 720,000 IU/kg every 8 hours for a maximum of 15 doses.

Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) and clinical laboratory evaluation 2 weeks after zanolimumab administration. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will be followed with this evaluation every 3-4 months until off study criteria are met.

If patients have stable disease or a partial response to treatment after the initial evaluation, or if a patient recurs or progresses after a clinical response, they may be eligible for re-treatment.

Patients will be entered into one of two strata: metastatic melanoma or metastatic renal cancer. Each of the strata will be conducted using an optimal two-stage phase II design to rule out an unacceptably low 15% clinical response rate, in favor of a modestly high response rate of 35% (p1=0.35).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Measurable metastatic melanoma or metastatic renal cancer. Metastatic cancer diagnosis will be confirmed by the Laboratory of Pathology at the National Cancer Institute (NCI).
* Patients must never have received high dose aldesleukin.
* Greater than or equal to 18 years of age.
* Willing to sign a durable power of attorney
* Able to understand and sign the Informed Consent Document
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Life expectancy of greater than three months.
* Patients of both genders must be willing to practice birth control for four months after receiving treatment.
* Serology:

  * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
  * Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the therapy on the fetus.
* Hematology:

  * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
  * White blood cell (WBC) (greater than 3000/mm^3).
  * Platelet count greater than 100,000/mm^3.
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
  * Serum creatinine less than or equal to 1.6 mg/dl.
  * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives zanolimumab, and patient's toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
* Six weeks must have elapsed since prior anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody therapy to allow antibody levels to decline, and patients who have previously received anti-CTLA4 antibody and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the therapy on the fetus or infant.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent systemic steroid therapy
* History of severe immediate hypersensitivity reaction to any of the agents used in this study. History of coronary revascularization or ischemic symptoms
* Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
* Documented LVEF of less than or equal to 45% tested in patients with:

  * History of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
  * Age greater than or equal to 60 years old.
* Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

  * A prolonged history of cigarette smoking (20 pack year of smoking within the past 2 years).
  * Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahmadzadeh M, Antony PA, Rosenberg SA. IL-2 and IL-15 each mediate de novo induction of FOXP3 expression in human tumor antigen-specific CD8 T cells. J Immunother. 2007 Apr;30(3):294-302. doi: 10.1097/CJI.0b013e3180336787. PMID 17414320
- [Background] Rosenberg SA. A new era for cancer immunotherapy based on the genes that encode cancer antigens. Immunity. 1999 Mar;10(3):281-7. doi: 10.1016/s1074-7613(00)80028-x. No abstract available. PMID 10204484
- [Background] Asano M, Toda M, Sakaguchi N, Sakaguchi S. Autoimmune disease as a consequence of developmental abnormality of a T cell subpopulation. J Exp Med. 1996 Aug 1;184(2):387-96. doi: 10.1084/jem.184.2.387. PMID 8760792

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HD IL-2 + Zanolimumab - Melanoma | HD IL-2 + Zanolimumab - Renal Cell
Started | 7 | 2
Completed | 7 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HD IL-2 + Zanolimumab - Melanoma | HD IL-2 + Zanolimumab - Renal Cell | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 8
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.9) | 61.0 (5.7) | 50.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 2 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Ability of a Combination of Aldesleukin (IL-2) and Zanolimumab (Anti-CD4 mAb) Administration to Mediate Tumor Regression in Patients With Metastatic Melanoma and Metastatic Kidney Cancer.
Description: Tumor regression was assessed by the Response Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% in the sum of the longest diameter (LD) recorded since the treatment started. Stable disease (SD) is neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD taking as reference the smallest sum LD.
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | HD IL-2 + Zanolimumab - Melanoma | HD IL-2 + Zanolimumab - Renal Cell
Number analyzed (Participants) | 7 | 2
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 0 | 0
  Progressive Disease | 7 | 2

2. Secondary Outcome: Toxicity of Zanolimumab and IL-2 Treatment Regimen
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 10 months
Measure: Number; unit: Participants
Arm/Group | HD IL-2 + Zanolimumab - Melanoma | HD IL-2 + Zanolimumab - Renal Cell
Number analyzed (Participants) | 7 | 2
Participants | 7 | 2

ADVERSE EVENTS:
Arm/Group | HD IL-2 + Zanolimumab - Melanoma | HD IL-2 + Zanolimumab - Renal Cell
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 7/7 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD IL-2 + Zanolimumab - Melanoma (N=7) | HD IL-2 + Zanolimumab - Renal Cell (N=2)
Hemoglobin (Blood and lymphatic system disorders) | 7 (14) | 2 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (7) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 7 (21) | 2 (5)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (6) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 6 (9) | 1 (3)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (3) | 0 (0)
Hypotension (Cardiac disorders) | 5 (8) | 2 (3)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 7 (14) | 2 (5)
Fatigue (General disorders) | 7 (17) | 2 (8)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 5 (12) | 2 (4)
Insomnia (General disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 6 (6) | 2 (2)
Sweating (diaphoresis) (General disorders) | 1 (1) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Hemorroids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (2)
Infection with unknown ANC (Infections and infestations) | 2 (5) | 0 (0)
Edema: limb (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (12) | 2 (7)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 6 (9) | 2 (4)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (15) | 2 (3)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (7) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 (12) | 1 (2)
Creatinine (Metabolism and nutrition disorders) | 4 (7) | 2 (4)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6 (15) | 2 (3)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (5) | 1 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (5) | 2 (4)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Mental status (Nervous system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (9) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Acute vascular leak syndrome (Vascular disorders) | 5 (8) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (3)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal-Other (Specify, upset stomach/gr 1) (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No